CLINICAL TRIAL: NCT04054336
Title: Mechanisms Underlying the Approach and Avoidance Task (AAT) in Alcoholic Inpatients
Brief Title: The Approach and Avoidance Task (AAT) in Alcoholic Inpatients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAT001
Record Dates: First submitted 2019-08-11; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Alcohol Dependence
Keywords: Approach and Avoidance Task, Inhibition
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Alcohol patients are randomly assigned to one of three conditions and are tested on three consecutive points in time.
Who Masked: Participant
Masking Description: Participants do not know that there exists more than one condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inhibition group (Experimental): The inhibition group gets the instructions to respond to pictures containing soft drinks by swiping/pulling them towards themselves, whereas pictures with alcoholic content shall be ignored. Up on pulling the pictures successively enlarge, whereas they shrink when ignored and slowly fade out.
  Interventions: Behavioral: Inhibit AAT
- Classical AAT group (Experimental): The classical AAT group is provided with a tablet on which an explicit AAT training is installed. Thus, just as participants in the inhibition group, participants are instructed to react upon soft drinks by swiping/pulling towards themselves the picture. Pictures containing alcoholic content shall be pushed away. Up on pulling pictures enlarge and up on pushing they shrink until they fade out.
  Interventions: Behavioral: classical AAT
- Control group (Sham Comparator): This type of active control group receives the instructions to swipe alcohol pictures to the left and soft drink pictures to the right (or vice versa depending on the sequential counterbalancing procedure).
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Inhibit AAT — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Inhibition group
Behavioral: classical AAT — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Classical AAT group
Behavioral: Control Group — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Control group

SUMMARY:
The approach and avoidance task (AAT) has evolved as a promising treatment add-on in the realm of psychology. Certain psychiatric diseases, such as behavioural addictions, social anxiety disorder, and arachnophobia, are characterized by a dysfunctional tendency to either approach or avoid disease-specific objects. This tendency can be measured by means of the approach and avoidance task. In this so-called diagnostic AAT participants are instructed to react upon the format or the frame colour of a picture. For instance, pictures have to be pushed away if they are presented in landscape format and pulled towards oneself if they are presented in portrait format (or vice versa). Hence, the format (or the frame colour) becomes the task-relevant dimension, whereas the content of the picture becomes the task-irrelevant dimension. However, what generally becomes obvious in the psychiatric diseases mentioned above is that the task-irrelevant dimension (picture content) exerts an influence on reaction times. For instance, alcoholic patients are generally faster to respond if alcoholic pictures are presented in a format requiring them to pull towards themselves and slower to respond if alcoholic pictures are shown in the format requiring them to push away a joystick. This behavioural tendency has been termed an approach bias for alcohol.

In order to counteract these dysfunctional approach or avoidance tendencies, an AAT-training has been developed. In this training participants/patients learn to either avoid or approach disease-specific objects. Alcohol-dependent patients, for instance, learn to avoid alcohol-related pictures by pushing or swiping the image away. It has been shown that these trainings can enhance treatment outcome (e.g. lower relapse rates) among alcohol-addicted patients (Wiers, Eberl, Rinck, Becker, & Lindenmeyer, 2011). The aim of the current study is to test whether the avoidance gesture is as important as suggested by the AAT's name or whether inhibiting the urge to approach alcoholic content might be enough to bring about the effect.

DETAILED DESCRIPTION:
The approach and avoidance task (AAT) has turned out as both a promising diagnostic tool as well as treatment add-on in psychological science. The AAT constitutes one form of cognitive bias modification (CBM), which has been shown to be particularly effective in the field of behavioral addictions, such as alcohol addiction (Eberl et al., 2013; Wiers et al., 2011). The general logic underlying the AAT is to carry out actions that are either compatible or incompatible with an individual's action tendencies. For instance, alcohol addicted patients tend to approach alcohol related stimuli faster than control pictures (i.e. soft drink stimuli), when they are instructed to react upon the format of a picture and not to its' content. This tendency of comparatively faster approaching and slower avoiding alcohol-related stimuli than soft drink content has been termed an approach bias for alcohol. The AAT as a therapeutic tool tries to counteract or at least to attenuate approach or avoidance biases by instructing patients to carry out approach and avoidance gestures that are in conflict with an individual's acquired action tendencies.

Whereas the general effectiveness of the AAT as a clinical intervention has been demonstrated several times, little is known about possible mechanisms that might subserve these effects. Therefore, the current study is dedicated to shed some light on one such potential mechanism, i.e. the role of the avoidance gesture within the alcohol-AAT.

As already suggested by the name of the AAT, the avoidance gesture seems to be a key ingredient in bringing about therapeutic effects. However, recent empirical evidence has brought about some interesting findings, giving rise to an alternative explanation.

A study by Kühn et al. (2017), contrary to common-held beliefs, indicated that inhibition capacity can be trained. Inhibition, in turn, consistently has been linked to psychopathology and all kinds of behavioural addictions (Smith, Mattick, Jamadar, & Iredale, 2014). The game by Kühn et al. (2017) used to train inhibition resembled the AAT in several ways, e.g. certain stimuli appearing on a treadmill had to be collected by swiping towards oneself and others had to be ignored and the objects slowly disappeared. The latter element contrasts with the AAT, since the ignored objects don't have to be pushed away. However, it resembles the AAT in the sense that in both cases stimuli slowly fade out of the screen and eventually disappear. These parallel let to the assumption that a new form of the alcohol AAT training might be equally effective in lowering relapse rates among alcoholic patients. More precisely, within the newly conceptualized AAT training patients are instructed to inhibit the urge to respond in response to alcohol-related content and to observe the stimuli fading out of the screen. In contrast, to the classical AAT training this zooming out of alcoholic stimuli is not conditional on an avoidance gesture, i.e. swiping/pushing away the stimulus.

It is hypothesized that compared to a control group, in which alcohol and soft drink stimuli have to be swiped to the left and right, both the classical AAT-and the inhibition group will show lower relapse rates and approach biases after the intervention, i.e. a training period of three weeks. No intergroup differences in terms of relapse rates and alcohol-related approach bias are expected for the classical AAT group and the inhibition group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol dependence (SKID-I)
* Abstinence from alcohol (at least 72 hours) and absence of major withdrawal symptoms
* Being in between 18-76 years of age
* Being able to understand rationales of the study and signing written informed consent
* Currently being inpatient seeking help overcoming alcohol dependence
* Medication allowed: Antiepileptic's (such as Carbamezepin), antidepressants, substances to treat other non-psychiatric diseases

Exclusion Criteria:

* Impaired ability to cooperate
* Presence of another substance dependency than alcohol and nicotine within the last year
* Presence of another axis-I disorder that interferes with the ability to cooperate within the study programme
* Current episode of a major depression
* Presence of axis-II disorders
* Presence of schizoaffective disorders
* Alcohol consumption in between withdrawal and start of the study
* Somatic or neurological disease that precludes the proper execution of the study
* Long-term intake of neuroleptics or hypnotics
* Current intake of benzodiazepines or Clomethiazol (in the period of five half-value times prior to the start of the study)
* Participation in other studies or other treatments than treatment as usual
* Planned long-term therapy after 3-week withdrawal programme
* Being homeless
* Prior electroconvulsive therapy
* Language barriers that preclude proper understanding of study contents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | 3 months
  Is measured by means of the timeline followback (TLFB). In the TLFB a thirty day period prior to hospitalization is inquired to get an impression of the alcohol consumption before detoxification. Both after the intervention period and at the follow-up measure 9 weeks after the end of the intervention period the TLFB is administered to the participants again. Thus, in total a period of 3 months after the enrollment in the study is captured by means of the TLFB and can be compared between groups and with baseline consumption of each individual.
Relapse rate | 3 months
  At each point of measurement it is inquired whether participants had a relapse. In order to enrich these self-reports, breathalysers are used to screen for possible alcohol intake prior to the appointment.

SECONDARY OUTCOMES:
Diagnostic AAT | 3 months
  In order to look whether participants' approach bias for alcohol changes as a consequence of the intervention, the diagnostic AAT is administered to all participants at every point of measurement.
Obsessive Compulsive Drinking Scale | 3 months
  A measure of aclohol addiction severity and craving.
Alcohol Urge Questionnaire | 3 months
  Assesses the urge to consume alcohol.
The State Trait Anxiety Inventory (STAI) | 3 months
  Is a commonly used measure of state and trait anxiety. Trait anxiety is assessed at the baseline measure, whereas potential changes in state anxiety are monitored across all three points of measurement of the study.
Positive and Negative Affect Schedule | 3 months
  Is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect.
Self-Control Scale | 3 months
  The self-control scale aims to assess people's ability to control their impulses, alter their emotions and thoughts, and to interrupt undesired behavioural tendencies and refrain from acting on them.
Becks's Depression Inventory | 3 months
  Assesses the degree of depressive symptoms.
Fagerström Test of Nicotine Dependence (FTND) | 3 months
  Fagerstrom test for nicotine addiction determines the degree of nicotine dependence based on smoking habits and frequency.
Barrett Impulsiveness Scale | 3 months
  A questionnaire designed to assess the personality/behavioral construct of impulsiveness.
Behavioral inhibition/avoidance scales | 3 months
  The BIS/BAS Scale is a 24-item self-report questionnaire designed to measure two motivational systems: the behavioral inhibition system (BIS), which corresponds to motivation to avoid aversive outcomes, and the behavioral activation system (BAS), which corresponds to motivation to approach goal-oriented outcomes.
Rating of pictures used in the study | 3 months
  Liking of all alcoholic and non alcoholic stimuli used in the study will be rated on a visual analogue scale, ranging from 0 to 100.
Expectancy Inventory of the intervention | 3 months
  Assesses an individual's expectancies and belief in positive outcomes associated with the training and alcohol treatment in general.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Kühn, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Clinic Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuhn S, Lorenz RC, Weichenberger M, Becker M, Haesner M, O'Sullivan J, Steinert A, Steinhagen-Thiessen E, Brandhorst S, Bremer T, Gallinat J. Taking control! Structural and behavioural plasticity in response to game-based inhibition training in older adults. Neuroimage. 2017 Aug 1;156:199-206. doi: 10.1016/j.neuroimage.2017.05.026. Epub 2017 May 17. PMID 28527788
- [Result] Eberl C, Wiers RW, Pawelczack S, Rinck M, Becker ES, Lindenmeyer J. Approach bias modification in alcohol dependence: do clinical effects replicate and for whom does it work best? Dev Cogn Neurosci. 2013 Apr;4:38-51. doi: 10.1016/j.dcn.2012.11.002. Epub 2012 Nov 14. PMID 23218805
- [Result] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Result] Smith JL, Mattick RP, Jamadar SD, Iredale JM. Deficits in behavioural inhibition in substance abuse and addiction: a meta-analysis. Drug Alcohol Depend. 2014 Dec 1;145:1-33. doi: 10.1016/j.drugalcdep.2014.08.009. Epub 2014 Aug 24. PMID 25195081